CLINICAL TRIAL: NCT03552614
Title: Movement Velocity and Fluidity Improve After Armeo®Spring Rehabilitation in Children Affected by Acquired and Congenital Brain Diseases: an Observational Study
Brief Title: Movement Improvement After Paediatric Armeo®Spring Rehabilitation
Status: Completed | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: Sol et Salus Hospital, Rimini, Italy (Unknown)
Responsible Party: Sponsor
Other Study IDs: 05/2018-Oss
Record Dates: First submitted 2018-05-30; First posted 2018-06-12 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Acquired Brain Injury; Cerebral Palsy
Keywords: robot-assisted rehabilitation; Armeo®Spring; quantitative assessment
MeSH Terms: conditions — Brain Injuries; Cerebral Palsy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- children with brain damage: Patients undergo physiotherapy + Upper limb robot-assisted rehabilitation
  Interventions: Device: Upper limb robot-assisted rehabilitation; Other: physiotherapy

INTERVENTIONS:
Device: Upper limb robot-assisted rehabilitation — Upper limb robot-assisted rehabilitation is performed with Armeo®Spring. It is a passive exoskeleton with five degrees of freedom that guarantees passive arm weight support with springs.
  The treatment was composed by 45 minutes of robotic training (5 times a week for 4 weeks) during which patients performed a customized pull of exergames.
  Other Names: Armeo Spring
Other: physiotherapy — Patients undergo 45-minute treatment sessions 5 times a week for 4 weeks of physiotherapy, focused on gross and fine motor ability to promote independence in daily activities, and it is customized on patients' need.

SUMMARY:
Children with acquired and congenital brain lesions (namely, cerebral palsy, CP, and acquired brain injury, ABI) may exhibit upper limb impairment, with consequent limitations in their daily living activities.

In recent years, robotic rehabilitation has become an important tool to promote functional recovery in patients with CP and ABI, thanks to its ability to promote high intensity, repetitive, engaging training. Moreover, it has additional advantages that can contribute to the understanding of the effectiveness of these devices in motor learning and recovery. It has indeed higher resolution and inter -rater and intra-rater reliability with respect to standard assessment methods (i.e. clinical scales). Furthermore, it is able to provide a quantitative evaluation of patients' movement during treatments instead of relying exclusively on qualitative observation. Recently, Merlo and co-workers (Sol et Salus, Rimini, Italy) developed and validated a tool to extract indices of accuracy, velocity and smoothness from the analysis of 3D trajectories of the end point of the robotic exoskeleton Armeo®Spring (Hocoma, CH).

The primary aim of the study is to retrospectively investigate the effectiveness of robot-assisted upper limb rehabilitation in children affected by congenital and acquired brain damages by means of funcional scales and quantitative assessment of movement performance (accuracy, velocity and smoothness).

Patients affected by acquired or congenital brain disease are enrolled. The inclusion criteria are: age between 5 and 18; the ability to handle objects in daily life within levels I, II, and III, according to the Manual Ability Classification System (MACS); the ability to understand and follow test instructions. Conversely, the exclusion criteria are: severe muscle contracture and/or spasticity, a diagnosis of severe learning disabilities or behavioral problems and visual or hearing difficulties that would impact on function and participation.

Participants undergo the standard intervention protocol followed at the IRCCS E. Medea. It is composed by 20 sessions with Armeo®Spring and 20 sessions of physiotherapy, within 1 month. Patients are evaluated before (T0) and after (T1) the intervention with the Quality of Upper Extremities Skills Test (QUEST) and the Melbourne Assessment of Unilateral Upper Limb Function. During the first, tenth and last training session, patients executed the "Vertical Capture" exergame, which assess patient's functional level during a task that involves elbow flex-extension and shoulder flex- extension and abd-adduction. From these evaluation sessions, quantitative indices of movement performance (precision, velocity and smoothness) are extracted.

ELIGIBILITY:
Inclusion Criteria:

* the ability to handle objects in daily life within levels I, II, and III, according to the Manual Ability Classification System (MACS);
* the ability to understand and follow test instructions.

Exclusion Criteria:

* severe muscle spasticity and/or contracture,
* diagnosis of severe learning disabilities or behavioral problems
* visual or hearing difficulties that would impact on function and participation

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Neurophysiatric care unit
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2018-05-20 (Actual); Study Completion 2018-05-20 (Actual)

PRIMARY OUTCOMES:
Quality of Upper Extremities Skills Test (QUEST) | baseline, after 1 month
  The QUEST is an internationally-validated scale that measures dissociated movement, grasp, weight-bearing and protective extension abilities in children with upper extremity movement disorders. The total score is the average of these four domain scores, with higher scores representing a better quality of movement.
Melbourne Assessment of Unilateral Upper Limb Function | baseline, after 1 month
  The Melbourne Assessment is a test that scores the quality of unilateral upper-limb motor function based on items involving reach, grasp, release and manipulation in neurologically impaired children
Hand Path Ratio (HPR) | baseline, after two weeks, after 1 month
  ratio between the pathway of the end effector and the straight trajectory between the initial and final positions of the end effector; the score is 100% for straight movements while it increases when curved trajectories are performed
horOS and verOS | baseline, after two weeks, after 1 month
  the horizontal and vertical overshooting of the movement (in cm) with respect to the target. It is a measure of the precision of the movement
velocity | baseline, after two weeks, after 1 month
  the mean and the maximum velocity of the 3D end-point trajectory (cm/s)
number of velocity peaks | baseline, after two weeks, after 1 month
  the number of peaks of the velocity profile. The lower is its value the smoother is the movement
normalized jerk | baseline, after two weeks, after 1 month
  computed as the differentiation of the 3D end-point trajectory. The lower is its value the smoother is the movement

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Biffi, PhD, Principal Investigator — Scientific Institute IRCCS E. Medea
Locations (1):
- Scientific Institute IRCCS E. Medea, Bosisio Parini, Lecco, Italy

REFERENCES:
- [Background] Frascarelli F, Masia L, Di Rosa G, Cappa P, Petrarca M, Castelli E, Krebs HI. The impact of robotic rehabilitation in children with acquired or congenital movement disorders. Eur J Phys Rehabil Med. 2009 Mar;45(1):135-41. PMID 19293759
- [Background] Turconi AC, Biffi E, Maghini C, Peri E, Servodio Iammarone F, Gagliardi C. Can new technologies improve upper limb performance in grown-up diplegic children? Eur J Phys Rehabil Med. 2016 Oct;52(5):672-681. Epub 2015 Nov 10. PMID 26554345
- [Background] Colombo R, Cusmano I, Sterpi I, Mazzone A, Delconte C, Pisano F. Test-retest reliability of robotic assessment measures for the evaluation of upper limb recovery. IEEE Trans Neural Syst Rehabil Eng. 2014 Sep;22(5):1020-9. doi: 10.1109/TNSRE.2014.2306571. Epub 2014 Feb 20. PMID 24760936
- [Background] Merlo A, Longhi M, Giannotti E, Prati P, Giacobbi M, Ruscelli E, Mancini A, Ottaviani M, Montanari L, Mazzoli D. Upper limb evaluation with robotic exoskeleton. Normative values for indices of accuracy, speed and smoothness. NeuroRehabilitation. 2013;33(4):523-30. doi: 10.3233/NRE-130998. PMID 24037096
- [Background] Longhi M, Merlo A, Prati P, Giacobbi M, Mazzoli D. Instrumental indices for upper limb function assessment in stroke patients: a validation study. J Neuroeng Rehabil. 2016 Jun 8;13(1):52. doi: 10.1186/s12984-016-0163-4. PMID 27278277